CLINICAL TRIAL: NCT02346942
Title: Factors Associated With Biologic Disease Modifying Antirheumatic Drugs Switching and Impact of Healthcare Resource Utilization in a Managed Care Setting
Brief Title: Factors Associated With Biologic DMARD Switching
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-474
Record Dates: First submitted 2014-09-29; First posted 2015-01-27 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients who have no history of bDMARD therapy use
- Patients who have a prior history of bDMARD therapy use

SUMMARY:
The Primary objective of this study is to understand the rheumatoid arthritis (RA) population in national integrated delivery network who are treated with first- or second-line biologic disease modifying anti-rheumatic drug (bDMARD) therapy (with or without Methotrexate) and to evaluate switching patterns and reasons for switching to another bDMARD.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Diagnosis of RA (ICD-9 714.xx) anytime during the study time period of 1/1/2007 to 10/31/2012
* Patients ≥18 years of age at diagnosis date
* Required to have to have 6 months pre-index and 12 months post-index continuous membership and drug benefit eligibility in the database

Exclusion Criteria:

* Patients less than 18 years of age on diagnosis date
* If they had a diagnosis of Crohn's disease, psoriasis, psoriatic arthritis, ulcerative colitis, ankylosing spondylitis, regional enteritis, or anal fistula during the pre-index period
* Patients who had <7 days supply of adalimumab or etanercept
* Patients currently in a clinical trial during our study
* If patients are in the second-line cohort and have more than 1 prior bDMARD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individual patients with RA will be identified using electronic medical records from 01/01/2007 to 10/31/2012. The medical file contains data on diagnostic and therapeutic services rendered in both inpatient and outpatient settings. The diagnoses and procedures for these services are coded using ICD-9-CM, Current Procedural Terminology (CPT), and Diagnosis-Related Group (DRG) codes with service dates.
Sampling Method: Non-Probability Sample
Enrollment: 4099 (Actual)
Dates: Start 2006-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Measure the change in population of patients who are treated with first- or second-line bDMARD therapy (with or without Methotrexate) to another bDMARD therapy | Approximately 12 months
  biologic disease modifying anti-rheumatic drug (bDMARD)
Measure the change in population of patients who are treated with first- or second-line bDMARD therapy (with or without Methotrexate) to another bDMARD therapy | Approximately 6 months
Measure the reasons for switching to another bDMARD based on Provider documentation in chart notes | 12 month post index follow up
Measure the reasons for switching to another bDMARD based on Provider documentation in chart notes | 6 months pre-index date

SECONDARY OUTCOMES:
Evaluate RA related and all cause healthcare resource utilization of doctor visits, hospitalizations and ER visits as patients switch bDMARDs measured from Patient heath claims data from KPSC integrated healthcare data | 6 month pre-index and 6 months pre-index date and 12 month post index follow up

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx